CLINICAL TRIAL: NCT00358501
Title: Defibrotide for the Treatment of Severe Hepatic Veno-Occlusive Disease in Hematopoetic Stem Cell Transplant Patients: A Historically-Controlled, Multi-Center Phase 3 Study to Determine Safety & Efficacy
Brief Title: Defibrotide for the Treatment of Severe Hepatic Veno-Occlusive Disease in Hematopoetic Stem Cell Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-01; NCT00410917 (obsolete NCT alias)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Severe Hepatic Veno-Occlusive Disease
Keywords: Defibrotide; Severe veno occlusive disease; Multi organ failure; Stem cell transplant; Liver; Regimen related toxicity; Day 100 survival
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease; Multiple Organ Failure | interventions — defibrotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Defibrotide (Experimental): Defibrotide treatment
  Interventions: Drug: Defibrotide
- Historical Control (No Intervention): Historical control group

INTERVENTIONS:
Drug: Defibrotide — Defibrotide 6.25 mg/kg i.v. administered four times a day via 2 hour continuous infusion. Minimum duration 21 days.
  Arms: Defibrotide

SUMMARY:
The purpose of this study is to (1) demonstrate the efficacy and safety (toxicity) of 25 mg/kg/day of Defibrotide in patients with severe veno-occlusive disease (sVOD) and (2) evaluate serum and endothelial markers of veno-occlusive disease (VOD) through the analysis of blood samples.

DETAILED DESCRIPTION:
This is a historically-controlled, multicenter, open label Phase 3 study to determine the safety and efficacy of 25 mg/kg/day of Defibrotide (DF) for the treatment of severe VOD in hematopoietic stem cell transplantation (HSCT) patients.

In this study, the term "severe VOD" is defined as those patients who meet the Baltimore diagnostic criteria for VOD (total bilirubin >/= 2.0 mg/dL plus two of the following: ascites, >/=5% weight gain and hepatomegaly), who also have multi-organ failure (i.e., pulmonary and/or renal dysfunction). This represents a group of patients in whom mortality at Day+100 has been estimated to be >80%.

Comparisons: The primary parameter is Complete Response at 100 days following stem cell transplant, utilizing historical controls as a comparator. The historical control database will be generated through a retrospective medical chart review performed at participating centers; the survival outcome of patients who would otherwise have met eligibility criteria for this trial will be compared to the survival observed in patients prospectively treated with Defibrotide. Secondary parameters include survival rate at 100 days and 6 months post stem cell transplantation (SCT), and special studies of endothelial and serum markers for VOD. This study will assess safety of the dose and schedule in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of VOD, defined by jaundice (bilirubin >/= 2 mg/dL) and at least 2 of the following clinical findings, by Day+21 post stem cell transplant: ascites; weight gain >/= 5% above baseline weight; hepatomegaly.
* Severe VOD, defined as VOD with multi-organ failure, i.e., presence of one or both of the following, by Day+28 post stem cell transplant: renal or pulmonary dysfunction.
* Provide voluntary written informed consent.

Exclusion Criteria:

* Pre-existing (prior to SCT) cirrhosis
* An alternative diagnosis for weight gain, ascites and jaundice
* Graft-versus-host disease (GVHD) grade B or higher involving liver or gut or grade C or higher involving skin
* Prior solid organ transplant
* Dependent on dialysis prior to and/or at the time of SCT
* Dependent on oxygen supplementation prior to SCT
* Significant acute bleeding or hemodynamic instability
* Requirement for the use of any medications that increase risk of hemorrhage will be excluded from the treatment group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (25):
- United States (22):
  - Duarte, California
  - Palo Alto, California
  - Denver, Colorado
  - Atlanta, Georgia
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Seattle, Washington
- Canada (3):
  - Vancouver, British Columbia
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Background] Richardson PG, Murakami C, Jin Z, Warren D, Momtaz P, Hoppensteadt D, Elias AD, Antin JH, Soiffer R, Spitzer T, Avigan D, Bearman SI, Martin PL, Kurtzberg J, Vredenburgh J, Chen AR, Arai S, Vogelsang G, McDonald GB, Guinan EC. Multi-institutional use of defibrotide in 88 patients after stem cell transplantation with severe veno-occlusive disease and multisystem organ failure: response without significant toxicity in a high-risk population and factors predictive of outcome. Blood. 2002 Dec 15;100(13):4337-43. doi: 10.1182/blood-2002-04-1216. Epub 2002 Aug 1. PMID 12393437
- [Background] Richardson, Soiffer, Antin, Voss, Jin, Kurtzberget al. Defibrotide (DF) for the Treatment of Severe Veno-Occlusive Disease (VOD) and Multi-System Organ Failure (MOF) Post SCT: Final Results of a Phase II, Multicenter, Randomized Study and Preliminary Analyses of Surrogate Markers and Ultrasound Findings. [abstract]. Blood. 2004;104 (11).
- [Derived] Richardson PG, Riches ML, Kernan NA, Brochstein JA, Mineishi S, Termuhlen AM, Arai S, Grupp SA, Guinan EC, Martin PL, Steinbach G, Krishnan A, Nemecek ER, Giralt S, Rodriguez T, Duerst R, Doyle J, Antin JH, Smith A, Lehmann L, Champlin R, Gillio A, Bajwa R, D'Agostino RB Sr, Massaro J, Warren D, Miloslavsky M, Hume RL, Iacobelli M, Nejadnik B, Hannah AL, Soiffer RJ. Phase 3 trial of defibrotide for the treatment of severe veno-occlusive disease and multi-organ failure. Blood. 2016 Mar 31;127(13):1656-65. doi: 10.1182/blood-2015-10-676924. Epub 2016 Jan 29. PMID 26825712
- See also: Click here for more information about Defibrotide. — http://www.gentium.com/Defibrotide.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Historical Control: The control group was selected from the historical medical charts of patients undergoing HSCT.
Period: Overall Study
Arm/Group | Defibrotide | Historical Control
Started | 102 | 32
Completed | 102 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Historical Control: The control group was selected from the historical medical charts of patients undergoing hematopoietic stem cell transplant (HSCT).
- Total: Total of all reporting groups
Arm/Group | Defibrotide | Historical Control | Total
Number analyzed (Participants) | 102 | 32 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (21.37) | 25.1 (20.23) | 25.7 (21.03)
Age, Customized [Number; unit: participants]
  ≤16 years old | 44 | 14 | 58
  >16 years old | 58 | 18 | 76
Gender [Count of Participants; unit: Participants]
  Female | 38 | 14 | 52
  Male | 64 | 18 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  White | 77 | 23 | 100
  Latino/Latina | 10 | 1 | 11
  African American | 6 | 2 | 8
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 4 | 10
  United States | 93 | 27 | 120
  Israel | 3 | 1 | 4
Weight [Mean (Standard Deviation); unit: kg] | 53.7 (33.73) | 52.6 (30.55) | 53.4 (32.89)

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day+100 Following Hematopoietic Stem Cell Transplant
Description: The 95.1% CI instead of 95% CI is used for the final analysis to provide a small adjustment for the fact that an interim analysis was performed.
Time Frame: Day+100 post hematopoietic stem cell transplant
Population: Intent-to-Treat
Measure: Number (95.1% Confidence Interval); unit: percentage of participants
Arm/Group | Defibrotide | Historical Control
Number analyzed (Participants) | 102 | 32
percentage of participants | 38.2 [28.8 to 47.7] | 25.0 [9.9 to 40.1]

2. Primary Outcome: Complete Response by Day+100 Post Hematopoietic Stem Cell Transplant
Description: as for outcome 1
Time Frame: Day+100 post hematopoietic stem cell transplant
Population: Intent-to-Treat
Measure: Number (95.1% Confidence Interval); unit: percentage of participants
Arm/Group | Defibrotide | Historical Control
Number analyzed (Participants) | 102 | 32
percentage of participants | 25.5 [17.0 to 34.0] | 12.5 [1.0 to 24.0]

3. Secondary Outcome: Survival at Day+180 Post Hematopoietic Stem Cell Transplantation
Description: as for outcome 1
Time Frame: 180 days post hematopoietic stem cell transplant
Population: Intent-to-Treat
Measure: Number (95.1% Confidence Interval); unit: percentage of participants
Arm/Group | Defibrotide | Historical Control
Number analyzed (Participants) | 102 | 32
percentage of participants | 32.4 [23.2 to 41.5] | 25.0 [9.9 to 40.1]

4. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events
Time Frame: Through 30 days from the last dose of Defibrotide
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Defibrotide | Historical Control
Number analyzed (Participants) | 102 | 32
percentage of participants
  Overall TEAEs | 97 | 100
  TEAEs that led to death | 64 | 69
  Treatment-emergent hemorrhage event | 64 | 75

5. Other Pre Specified Outcome: Historical Control Group Adverse Event Information
Description: Historical Control group was not assessed for severity
Time Frame: Through 30 days from the last dose of Defibrotide
Measure: Number; unit: Number of patients
Arm/Group | Historical Control
Number analyzed (Participants) | 32
Number of patients
  Total Number of Participants Affected | 32
  Coagulopathy | 5
  Anaemia | 1
  Disseminated intravascular coagulation | 1
  Thrombocytopenia | 1
  Haemorrhagic anaemia | 1
  Tachycardia | 14
  Bradycardia | 6
  Cardiac arrest | 2
  Atrial fibrillation | 1
  Cardiac failure congestive | 2
  Sinus tachycardia | 1
  Cardio-respiratory arrest | 1
  Ventricular tachycardia | 1
  Acute myocardial infarction | 1
  Cardiac failure | 1
  Cardiac tamponade | 1
  Dilatation ventricular | 1
  Pericarditis uraemic | 1
  Supraventricular tachycardia | 1
  Systolic dysfunction | 1
  Tachyarrhythmia | 1
  Ventricular hypokinesia | 1
  Adrenal haemorrhage | 1
  Euthyroid sick syndrome | 1
  Conjunctival haemorrhage | 3
  Ocular icterus | 1
  Scleral haemorrhage | 1
  Conjunctival hyperaemia | 1
  Dry eye | 1
  Eye discharge | 1
  Eye haemorrhage | 1
  Eye irritation | 1
  Lid sulcus deepened | 1
  Pupils unequal | 1
  Diarrhoea | 12
  Vomiting | 8
  Nausea | 10
  Abdominal pain | 7
  Constipation | 5
  Gastrointestinal haemorrhage | 3
  Haematemesis | 3
  Lip haemorrhage | 4
  Mouth haemorrhage | 3
  Dyspepsia | 1
  Haematochezia | 3
  Melaena | 2
  Retching | 1
  Abdominal distension | 1
  Chapped lips | 1
  Gastrointestinal hypomotility | 2
  Gastrointestinal sounds abnormal | 1
  Upper gastrointestinal haemorrhage | 1
  Abdominal discomfort | 1
  Abdominal tenderness | 1
  Duodenal perforation | 1
  Duodenal ulcer | 1
  Dysphagia | 1
  Epigastric discomfort | 1
  Gastritis | 1
  Lip swelling | 1
  Lower gastrointestinal haemorrhage | 1
  Oesophagitis | 1
  Oral disorder | 1
  Pancreatitis | 1
  Umbilical hernia | 1
  Pyrexia | 9
  Multi-organ failure | 3
  Oedema peripheral | 4
  Generalised oedema | 8
  Hypothermia | 5
  Oedema | 7
  Pain | 3
  Face oedema | 3
  Asthenia | 1
  Chills | 2
  Catheter site erythema | 1
  Irritability | 2
  Catheter site swelling | 1
  Systemic inflammatory response syndrome | 1
  Thrombosis in device | 1
  Catheter site related reaction | 1
  Extravasation | 1
  Polyserositis | 1
  Venoocclusive liver disease | 2
  Hepatic failure | 3
  Jaundice | 3
  Hepatorenal syndrome | 2
  Acute hepatic failure | 1
  Cholelithiasis | 1
  Gallbladder disorder | 1
  Hepatomegaly | 1
  Portal vein thrombosis | 1
  Graft versus host disease in skin | 5
  Graft versus host disease | 2
  Graft versus host disease in intestine | 2
  Graft versus host disease in liver | 3
  Engraftment syndrome | 1
  Hypogammaglobulinaemia | 1
  Sepsis | 2
  Septic shock | 2
  Bacteraemia | 3
  Cytomegalovirus infection | 1
  Pneumonia | 1
  Candida sepsis | 1
  Candidiasis | 1
  Enterococcal infection | 1
  Catheter site infection | 1
  Enterococcal sepsis | 1
  Oral candidiasis | 1
  Sinusitis | 2
  Staphylococcal bacteraemia | 1
  Bacterial infection | 1
  Clostridium difficile colitis | 1
  Herpes simplex | 1
  Nasopharyngitis | 1
  Osteomyelitis chronic | 1
  Pneumonia fungal | 1
  Streptococcal bacteraemia | 1
  Urinary tract infection enterococcal | 1
  Vaginal infection | 1
  Post procedural haemorrhage | 1
  Contusion | 2
  Laceration | 1
  Periorbital haemorrhage | 2
  Toxicity to various agents | 2
  Periorbital contusion | 1
  Endotracheal intubation complication | 1
  Eschar | 1
  Eye contusion | 1
  Scratch | 1
  Wound haemorrhage | 1
  Wound secretion | 1
  Blood urine present | 2
  Haematocrit decreased | 2
  Heart rate increased | 1
  Activated partial thromboplastin time prolonged | 1
  Ammonia increased | 1
  Blood urea increased | 1
  Blood urine | 1
  Breath sounds abnormal | 1
  Cardiac murmur | 1
  Haemoglobin decreased | 1
  Occult blood positive | 1
  Prothrombin time prolonged | 1
  Transaminases increased | 1
  Urine output decreased | 1
  Hyperglycaemia | 4
  Fluid overload | 5
  Metabolic acidosis | 4
  Hypovolaemia | 2
  Acidosis | 2
  Decreased appetite | 1
  Hypercalcaemia | 1
  Hypernatraemia | 1
  Fluid retention | 1
  Hypervolaemia | 1
  Hypoalbuminaemia | 1
  Lactic acidosis | 1
  Type 2 diabetes mellitus | 1
  Back pain | 3
  Muscle spasms | 1
  Myalgia | 1
  Groin pain | 1
  Limb discomfort | 1
  Pain in extremity | 1
  Pain in jaw | 1
  Convulsion | 3
  Tremor | 4
  Cerebral haemorrhage | 1
  Somnolence | 2
  Asterixis | 1
  Lethargy | 1
  Mental impairment | 1
  Brain oedema | 1
  Paralysis | 1
  Intercranial pressure increased | 1
  Peripheral nerve palsy | 1
  Agitation | 9
  Confusional state | 5
  Anxiety | 4
  Mental status change | 1
  Insomnia | 4
  Depression | 1
  Disorientation | 4
  Paranoia | 1
  Haematuria | 5
  Cystitis haemorrhagic | 1
  Renal failure | 1
  Bladder spasm | 3
  Incontinence | 2
  Anuria | 1
  Azotaemia | 1
  Bladder outlet obstruction | 1
  Chromaturia | 1
  Pollakiuria | 1
  Urinary retention | 1
  Scrotal oedema | 2
  Oedema genital | 1
  Perineal pain | 1
  Vaginal haemorrhage | 1
  Vulvovaginal erythema | 1
  Epistaxis | 5
  Pulmonary alveolar haemorrhage | 5
  Respiratory failure | 4
  Pleural effusion | 6
  Cough | 3
  Rales | 6
  Dyspnoea | 5
  Tachypnoea | 2
  Apnoea | 1
  Atelectasis | 2
  Nasal flaring | 3
  Oropharyngeal pain | 1
  Acute respiratory distress syndrome | 1
  Haemothorax | 1
  Pneumonia aspiration | 2
  Respiratory distress | 2
  Sputum discoloured | 1
  Wheezing | 1
  Bronchial haemorrhage | 1
  Bronchial secretion retention | 1
  Haemoptysis | 1
  Hyperventilation | 1
  Idiopathic pneumonia syndrome | 1
  Pneumomediastinum | 1
  Pneumonitis | 1
  Pulmonary embolism | 1
  Respiratory acidosis | 1
  Respiratory disorder | 1
  Respiratory tract oedema | 1
  Upper respiratory tract congestion | 1
  Use of accessory respiratory muscles | 1
  Petechiae | 9
  Rash | 7
  Blister | 8
  Decubitus ulcer | 1
  Erythema | 3
  Pruritus | 3
  Skin disorder | 5
  Alopecia | 5
  Rash erythematous | 2
  Ecchymosis | 1
  Skin ulcer | 2
  Blood blister | 1
  Skin exfoliation | 2
  Dermatitis bullous | 1
  Purpura | 1
  Rash macular | 1
  Generalised erythema | 1
  Hyperhidrosis | 1
  Rash maculo-papular | 1
  Skin discolouration | 1
  Skin hypopigmentation | 1
  Skin necrosis | 1
  Hypotension | 16
  Capillary leak syndrome | 2
  Ischaemia | 1
  Pallor | 1
  Circulatory collapse | 1
  Hypertension | 1
  Hypovolaemic shock | 1
  Shock | 1

ADVERSE EVENTS:
Description: All adverse events data for Historical Control is provided as an Outcome Measure. Historical Control group summary adverse event information is only available without severity and therefore indicated as 0 at risk in the adverse event tables.
Arm/Group | Defibrotide | Historical Control
Serious Adverse Events (participants affected / at risk) | 80/102 | 0/0
Other Adverse Events (participants affected / at risk) | 91/102 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=102) | Historical Control (N=0)
Thrombotic thrombocytopenia purpura (Blood and lymphatic system disorders) | 3 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 0
Multi-organ failure (General disorders) | 15 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 10 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 0
Sepsis (Infections and infestations) | 6 | 0
Septic shock (Infections and infestations) | 3 | 0
Intracranial hemorrhage (Nervous system disorders) | 4 | 0
Cerebral hemorrhage (Nervous system disorders) | 3 | 0
Renal failure (Renal and urinary disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Pulmonary alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hypotension (Vascular disorders) | 14 | 0
Coagulopathy (Blood and lymphatic system disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Tay-Sachs disease (Congenital, familial and genetic disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 2 | 0
Puncture site haemorrhage (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Systematic inflammatory response syndrome (General disorders) | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Liver disease (Hepatobiliary disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 2 | 0
Graft versus host disease in skin (Immune system disorders) | 1 | 0
Candida sepsis (Infections and infestations) | 2 | 0
Enterococcal infection (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Human herpes virus 6 serology (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide (N=102) | Historical Control (N=0)
Hypotension (Vascular disorders) | 31 | 0
Diarrhea (Gastrointestinal disorders) | 24 | 0
Vomiting (Gastrointestinal disorders) | 20 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 0
Nausea (Gastrointestinal disorders) | 13 | 0
Pyrexia (General disorders) | 14 | 0
Bradycardia (Cardiac disorders) | 9 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 10 | 0
Haematuria (Renal and urinary disorders) | 10 | 0
Tachycardia (Cardiac disorders) | 10 | 0
Catheter site hemorrhage (General disorders) | 7 | 0
Conjunctival hemorrhage (Eye disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Generalized edema (General disorders) | 8 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 0
Mental status change (Psychiatric disorders) | 7 | 0
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 6 | 0
Blister (Skin and subcutaneous tissue disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 6 | 0
Headache (Nervous system disorders) | 6 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 0
Oedema peripheral (General disorders) | 13 | 0
Agitation (Psychiatric disorders) | 11 | 0

LIMITATIONS AND CAVEATS:
Primary endpoint was changed after all patients were treated and current results reflect the final protocol. Adverse event severity was only reported for treatment group as control group was not assessed for severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No